CLINICAL TRIAL: NCT06801210
Title: The Weight of Victory: Exploring Short- and Long-term Health Outcomes in Former Male & Female Elite Atheltes from Weight-sensitive Sports
Brief Title: The Weight of Victory: Exploring Short- and Long-term Health Outcomes in Former Male & Female Elite Athletes from Weight-sensitive Sports
Status: Not yet recruiting | Type: Observational
Sponsor: Norwegian School of Sport Sciences (Other)
Responsible Party: Principal Investigator, Professor Jorunn Sundgot-Borgen, Professor, Norwegian School of Sport Sciences
Other Study IDs: 841008
Record Dates: First submitted 2025-01-16; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Musculoskeletal Health; Fertility; Mental Health; Quality of Life; Body Image; Disordered Eating
Keywords: Elite athletes; Mental health; Somatic health; Disordered eating; Musculoskeletal health; Quality of life; Anxiety and depression; Behavioral; Reproductive health; Fertility; Harassment; Body acceptance; Personality traits; Weight regulation
MeSH Terms: conditions — Psychological Well-Being; Anxiety Disorders; Depression; Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

GROUPS / COHORTS (3):
- Former elite athletes from weight-sensitive sports: Former elite athletes from weight-sensitive sports. Including former elite athletes from weight-class, gravitational, aesthetic, and certain endurance type of sports.
- Former elite athletes from less weight-sensitive sports: Former elite athletes from less weight-sensitive sports. Including team sports (e.g. handball, soccer, basketball)
- General population: An age matched reference group for the groups of former elite athletes. Includes a sample from the general population without a background as an elite athlete.

SUMMARY:
The health of former elite athletes has been identified as a critical research gap where there is limited knowledge about both short- and long-term consequences after ending their careers. The transition phase from an active elite career to everyday life has been shown to be particularly problematic, yet this issue has been little studied among former Norwegian elite athletes. Furthermore, questions remain regarding the health of athletes from weight-sensitive sports, such as weight-class, aesthetic, and certain endurance sports. These athletes face specific challenges related to maintaining a certain physique and frequent changes in body weight during their active careers. This group has been shown to be vulnerable to a range of problematic health outcomes related to low energy availability, and little is known about the long-term effects of a career involving this.

Therefore, the overall purpose of the project is to map the mental and physical health of former elite athletes. At the same time, there will be a particular focus on the differences between weight-sensitive and less weight-sensitive sports, different types of sports, gender, as well as previous dieting and eating behaviors.

DETAILED DESCRIPTION:
The project will be a quantitative cross-sectional study that includes former elite athletes from both weight-sensitive and less weight-sensitive sports, as well as a sample from the general population for comparison. Information will be collected via an electronic questionnaire that surveys a range of physical and mental health variables among the participants. In addition, behavioral variables related to impulse control, eating and dieting patterns, and weight regulation will be assessed.

Furthermore, the project is expected to contribute new knowledge by identifying health challenges and the explanatory variables for these challenges among former elite athletes. Thus, the project can inform the development of targeted preventive measures, interventions, and policy changes that can improve health and quality of life both during and after athletes' careers and be of significant importance for future athletes.

ELIGIBILITY:
Inclusion Criteria:

* Represented the national team at senior and/or junior level, (Non-organized sports) competed at national and/or international level. , >1 year since retirement , >18 years old,and a proficient level of Norwegian reading and writing skills

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Former male and female Norwegian elite athletes and a age matched controls from the general population
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-01-30 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Symptoms of eating disorders (Eating Disorder Examination Questionnaire, EDE-Q) | January 2025 to June 2025
  This outcome measure will use the Eating Disorder Examination Questionnaire (EDE-Q) to assess the frequency and severity of eating disorder symptoms. The EDE-Q is a validated self-report questionnaire covering dietary restraint, eating concern, shape concern, and weight concern
Pain, function, and overall well-being connected to musculoskeletal status (Musculoskeletal Health Questionnaire, MSK-HQ) | From January 2025 to June 2025
  This outcome measure will use the Musculoskeletal Health Questionnaire (MSK-HQ) to assess self-reported musculoskeletal health. The MSK-HQ is a validated instrument covering key domains such as pain, function, and overall well-being in individuals with musculoskeletal conditions. It provides a comprehensive overview of the patient's musculoskeletal status, including symptoms and the impact on daily activities.
Menstrual function and history & fertility function and history (The Low Energy Availability in Males Questionnaire, LEAM-Q, Low Energy Availability in Females Questionnaire, LEAF-Q, and The Norwegian Mother, Father and Child Cohort Study, MoBa) | From January 2025 to June 2025
  Items from The validated Low Energy Availability in Females Questionnaire (LEAF-Q) will be included to assess menstrual function (Melin et al., 2014). Items from The Low Energy Availability in Males Questionnaire (LEAM-Q) (Lundy et al., 2022) will be included for assessing reproductive health among the male participants. In addition, questions from The Norwegian Mother, Father and Child Cohort Study (MoBa) will be included to cover fertility status.

SECONDARY OUTCOMES:
Symptoms of Psychological Distress (Symptom Checklist-10, SCL-10) | From January 2025 to June 2025
  This outcome measure will use the Symptom Checklist-10 (SCL-10) to assess the frequency and severity of common mental distress symptoms. The SCL-10 is a validated, abbreviated version of the SCL family of instruments (e.g., SCL-25, SCL-90) that covers core areas such as anxiety, depression, and somatic complaints. It provides an overall indication of the level of psychological distress and can be used for both screening and monitoring changes over time.
Alchohol and drug use (Alcohol Use Disorders Identification Test - Consumption, AUDIT-C and Drug Use Disorders Identification Test, DUDIT) | From January 2025 to June 2025
  The AUDIT-C assesses alcohol consumption, drinking behaviors, and alcohol-related issues (Babor et al., 2001). The Drug Use Disorders Identification Test (DUDIT) will be included. The DUDIT assesses symptoms of substance abuse, as well as harmful use, and drug dependence.
Satisfaction With Life (Satisfaction With Life Scale, SWLS) | From January 2025 to June 2025
  This outcome measure will use the Satisfaction With Life Scale (SWLS) to evaluate individuals' overall assessments of their own life satisfaction. The SWLS is a validated, brief questionnaire comprising five statements that respondents rate based on their level of agreement. It captures the cognitive judgment of one's life quality, providing a reliable indicator of subjective well-being and overall life satisfaction.
Cognitive Function (PROMIS® v2.0 Cognitive Function-Short Form 6a) | From January 2025 to June 2025
  This outcome measure will utilize the PROMIS® v2.0 Cognitive Function-Short Form 6a to assess individuals' self-reported cognitive abilities. The PROMIS Cognitive Function-Short Form 6a is a validated, brief questionnaire designed to evaluate various aspects of cognitive performance, including memory, concentration, and mental clarity
Body Appreciation and Muscle Dysmorphic Disorder Symptoms (Body Appreciation Scale-2, BAS-2, and the Muscle Dysmorphic Disorder Inventory, MDDI) | From January 2025 to June 2025
  The Body appreciation scale-2 (BAS-2) is a 10-item measure of an individual's acceptance, opinions and respect of their own body, The questionnaire is validated. Body satisfaction will be measured with the inclusion of the Muscle Dysmorphic Disorder Inventory (MDDI). The MDDI is a 13-item self-report measure which have three sub-scales assessing clinical features associated with muscle dysmorphia (MD), including drive for size, functional impairment, and appearance intolerance

OTHER OUTCOMES:
Experiences of harassment, maltreatment, and abuse. | From January 2025 to June 2025
  To assess harassment, maltreatment and abuse a modified version of the questionnaire developed by Sølvberg et al (2022) will be included. This version will include questions regarding the participants experiences with harassment in their active career, and will include questions on physical, psychological, sexual (contact and non-contact), and neglecting harassment and/or abuse.
  Reference:
  Sølvberg N, Torstveit MK, Rosenvinge JH, Pettersen G, Sundgot-Borgen J. Sexual Harassment and Abuse among Young Elite Athletes, Recreational Athletes, and Reference Students: A Prospective Study. Med Sci Sports Exerc. 2022 Nov 1;54(11):1869-1878. doi: 10.1249/MSS.0000000000002972. Epub 2022 Jun 24. PMID: 35763597; PMCID: PMC9584052.

IPD SHARING:
Plan to Share IPD: Undecided